CLINICAL TRIAL: NCT01832545
Title: The PICO Project: Aquatic Exercise for Knee Osteoarthritis in Overweight and Obese Individuals
Brief Title: Aquatic Exercise Program for Knee Osteoarthritis
Acronym: PICO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Lisbon (Other)
Responsible Party: Principal Investigator, Flávia Yázigi, Master Degree in Exercise and Health, PhD student (credits concluded); Professor assistent;, Technical University of Lisbon
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PICO-FY013
Record Dates: First submitted 2013-04-10; First posted 2013-04-16 (Estimated); Last update posted 2013-04-16 (Estimated); Status verified 2013-04

CONDITIONS: Knee Osteoarthritis; Obesity
Keywords: Aquatic exercise; Knee Osteoarthritis; Exercise; Pain; Obesity.
MeSH Terms: conditions — Osteoarthritis, Knee; Obesity; Motor Activity; Pain | interventions — Aquatic Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Educational Program (Active Comparator): The communitarian PESO program is based on appropriate clinical guidelines and on validated behavior change principles. Implemented by an intervention team with expertise gained from current scientific research in weight control determinants, this program as well PICO, is free of charge for all interested adults who wish to manage their weight and health. It operates since 2005 with the aims to prevent obesity or reduce excess weight, as well as, some of the risks associated with obesity in adults through a change to steady healthy habits, attitudes and behaviors. PESO has 3 months duration and it is structured in 12 sessions of one and a half hour, once a week.
  Interventions: Behavioral: Educational Program
- Aquatic Exetcise (Experimental): Aquatic Exercise program is organized in 24 sessions distributed over 12 consecutive weeks, with a frequency of twice a week. The duration of each session will be 60 minutes, being that 10 minutes are for patient reception, blood pressure control, pain register or others and the effective time inside the water is 45 minutes. The indoor pool works with an air temperature around 27±1ºC and water temperature is controlled for 30.5±5ºC. Workout is organized in order to have a progressive overload every week or every two sessions, when occurs an introduction of a new stimulus. Water is the main instrument to create resistance and only in the last weeks, according with participants progression and if the self-reported pain controlled, drag equipment will be added.
  Interventions: Other: Aquatic Exercise

INTERVENTIONS:
Other: Aquatic Exercise
  Arms: Aquatic Exetcise
Behavioral: Educational Program — Control Group
  Arms: Educational Program

SUMMARY:
The aim of PICO study is to design an aquatic exercise program specific for obese individuals with knee osteoarthritis which the main goals are OA symptoms management and the improvement of physical fitness. The author's opinion is that the musculoskeletal pain is the main constraint for any kind of mobility and its control should be considered as an important goal in the weight management's programs. Therefore the PICO project proposes an aquatic exercise program to controlling pain and other symptoms management, showing that it is possible to live with the disease, and motivating the change in lifestyle, thus preventing the installation or worsening of KOA. In this way, five hypotheses were formulated: H1. 3 months of aquatic exercise is enough to improve KOA symptoms and functionality in obese individuals; H2. The gait parameters of obese individuals with KOA can be improved by aquatic exercise; H3. Beyond the exercises skills, aquatic exercise group classes can work with an educational component, promoting lifestyles changes. H4: Pain reduction and a better psychological status can lead an increase of functionally, increasing amount of physical activity. H5: Even if the main goal is not weight management, the aquatic exercise program can lead a weight reduction or body composition change.

DETAILED DESCRIPTION:
The PICO program is an overall body fitness and mind intervention through aquatic exercise involving as well an education component, created specifically for individuals with KOA. Its a single-blinded, one center, and randomized controlled trial with 3 months duration. Participants will be randomized into one of two groups: aquatic exercise (AE) and control group (CG) which will participate in an educational program with the same hourly load.

ELIGIBILITY:
Inclusion Criteria:

* The study sample will consist of 60 adults, community-dwelling (Lisbon) people with: (1) age 40-65 years; (2) 28.0 ≤ BMI ≤ 45 kg/m2; unilateral or bilateral KOA (3) knee pain (4) grade I-III radiographic tibiofemoral OA or tibiofemoral plus patellofemoral OA (5) a sedentary lifestyle, defined as not participating in a program that incorporates more than 30 minutes per week of formal exercise within the past 6 months; (6) being independent with mobility capacity; and (7) reading and writing knowledge.

Exclusion Criteria:

* Subjects with skin diseases, unstable medical conditions and with hip or knee replacement, knee surgery within the past 6 months and participants who had any type of knee injections within the past 3 months will be excluded of PICO.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-11; Primary Completion 2012-04 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Knee Osteoarthritis symptoms | "Change" (e.g., "baseline and 12 weeks")
  Pain, stiffness and other symptoms should be assessed by the Brief Pain Inventory (BPI); Numerical Rating Scale (NRS) and by the Knee Injury and arthritis Outcome Score (KOOS)
Health Quality of Life | "Change" (e.g., "baseline and 12 weeks")
  The MOS Short-Form Health Survey (SF-12)and the Beck Depression Inventory (BDI-II) will be used to asses Quality of life and Psychological status
Physical Function | "Change" (e.g., "baseline and 12 weeks")
  Physical function will be assessed by the following functional tests: The Six Minutes Walking Test to verify aerobic capacity and the walking ability; The Chair Sit and Reach test for hamstring flexibility; The Back Scratch Test for overall shoulder range of motion; The Five-Repetition Sit-To-Stand Test for functional strength .
Strength | "Change" (e.g., "baseline and 12 weeks")
  A dynamometer will be used for isokinetic assessment of knee strength (flexor and extensor muscles) and isometric knee strength, bilaterally; The Handgrip Strength Test will evaluate maximal isometric force of the muscles of the hand and forearm.
Gait | "Change" (e.g., "baseline and 12 weeks")
  Kinematics and kinetics outcomes will be analyzed from gait test (gait speed, gait cycle, ground reaction forces and knee forces moments).

SECONDARY OUTCOMES:
Body composition | "Change" (e.g., "baseline and 12 weeks")
  Body composition. Body Mass Index and a dual energy x-ray absorptiometry (DXA) scanner will be used to measure whole body lean mass, fat mass and bone mineral content.
Body Morphology | "Change" (e.g., "baseline and 12 weeks")
  Body Morphology will be registered by anthropometric measurements (body mass, stature, foot length, and waist, hip, mid-thigh and calf circumference).
Lifestyle | "Change" (e.g., "baseline and 12 weeks")
  Lifestyle should be assessed by International Physical Activity Questionnaire (IPAQ)and by the Weight and Lifestyle Inventory (WALI).
Inflammatory Markers | "Change" (e.g., "baseline and 12 weeks")
  The main measures are Interleukin 6 (IL-6),high-sensitivity C-reactive protein (HsCRP), TNFα and TNFα soluble receptor 1(sTNFR1).

CONTACTS AND LOCATIONS:
Overall Officials: Margarida Espanha, PhD, Study Chair — Technical University of Lisbon
Locations (1):
- Technical University of Lisbon, Lisbon, Cruz Quebrada-Dafundo, Portugal

REFERENCES:
- [Derived] Yazigi F, Espanha M, Marques A, Teles J, Teixeira P. Predictors of walking capacity in obese adults with knee osteoarthritis. Acta Reumatol Port. 2018 Oct-Dec;43(4):256-263. PMID 30641533
- [Derived] Yazigi F, Espanha M, Vieira F, Messier SP, Monteiro C, Veloso AP. The PICO project: aquatic exercise for knee osteoarthritis in overweight and obese individuals. BMC Musculoskelet Disord. 2013 Nov 13;14:320. doi: 10.1186/1471-2474-14-320. PMID 24219758